CLINICAL TRIAL: NCT03847623
Title: Effect of Preoperative Curcumin in Breast Cancer Patients
Acronym: EPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Nur Aishah Mohd Taib, Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20149-582
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin (Experimental): Capsules, taken orally, 8g per day (Bi-daily dosing)
  Interventions: Dietary Supplement: Curcumin
- Placebo (Placebo Comparator): Capsules, taken orally, bi-daily dosing
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — Natural compound, active ingredient of turmeric, in bi-daily dosing
  Arms: Curcumin
Other: Placebo — Placebo tablets at bi-daily dosing
  Arms: Placebo

SUMMARY:
Effect of curcumin on modulation of immune and inflammatory parameters in pre-operative patients

DETAILED DESCRIPTION:
Patients diagnosed with breast cancer will be supplemented with either curcumin or placebo for a minimum period of 2 weeks and may be extended up to 4 weeks prior to their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with operable breast cancer
* Life expectancy of at least 3 months
* Adequate organ function
* No allergy to curcumin
* Provides consent to participate in trial and adhere to the study protocol

Exclusion Criteria:

* Receiving concomitant radiotherapy, hormonal, immune therapy or other investigational drugs
* Uncontrolled concurrent illness
* Patient of anti platelet medications
* Pregnant / breast feeding
* Patients who are unable or unwilling to take curcumin, herbal remedies, or non-prescription medications
* Patients with bleeding tendency, bleeding disorders and abnormal bleeding/clotting profile

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumour infiltrating lymphocytes (TILs) | For 2 to 4 weeks
  Scoring as per recommendations by International Immuno-Oncology Biomarker Working Group

SECONDARY OUTCOMES:
FOXP3 | For 2 to 4 weeks
  Immunohistochemistry analysis
CD68 | For 2 to 4 weeks
  Immunohistochemistry analysis

CONTACTS AND LOCATIONS:
Overall Officials: Nur Aishah Taib, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Malaysia